CLINICAL TRIAL: NCT04798170
Title: Fetal Nasal Bone Length Nomogram at 11-13wk+6 Days in Upper Egyptain Pregnant Women
Brief Title: Fetal Nasal Bone Length Nomogram at 11-13wk+6days in Upper Egyptian Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, mostafa mahmoud hassan mohamed, Sohag, Sohag University
Other Study IDs: Soh-Med-21-03-05
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Nasal Bone Length

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Utrasound — Ultrasound examination

SUMMARY:
establish a reference values for the fetal nasal bone length (NBL) in upper egyptian pregnant women at 11-13wk+6 days

DETAILED DESCRIPTION:
By using ultrasound measure fetal nasal bone length at 11-13wk+6days in Upper Egyptian pregnant women in mid-sagittal view in single pregnancy

ELIGIBILITY:
Inclusion Criteria:

Normal antenatal women of gestational age between 11 to 13week +6days. Single pregnancy. Viable fetus. No fetal malformation. No previous history of fetal malformation

Exclusion Criteria:

Medical diseased women . Multiple gestations . Fetal malformations . Missed abortion .

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Non diseased Pregnant women at 11-13wk+6 days of gestation in single pregnancy without previous history of congenital anomalies
Study Population: Cross sectional study of pregnant women in Upper Egypt at 11-13wk of gestation
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Fetal nasal bone length nomogram | 2 years
  Establish nomogram for nasal bone length in Upper Egyptian pregnant women